CLINICAL TRIAL: NCT06197867
Title: Prevalence of Metabolic Liver Disorders in Children Attending Gastroenterology and Hepatology Unit at Assuit University Children Hospital.
Brief Title: The Prevalence of Metabolic Liver Disorders in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Beshoi Markos Moner Mashreky, Assiut university, Assiut University
Other Study IDs: Metabolic liver disorders
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Metabolic Liver Disorders in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of study :

To detect the prevalence of metabolic liver disease in patients attending gastroenterology and hepatology unit at assuit university children hospital.

DETAILED DESCRIPTION:
Metabolic Liver Disease is a group of metabolic disorders that stops the liver to function or fail. These metabolic conditions affect the pathways in the liver cells - the pathways that help the body break down, absorb, process, transport, and store nutrients like amino acids, carbohydrates and fats.

Metabolic liver diseases (MLD), an inborn error of metabolism, is caused by defect of single enzyme or transport protein resulting into abnormality in synthesis or catabolism of carbohydrate, protein and fat.

The pathogenesis of MLD can be divided into three groups:

1. Defect in the intermediary metabolic pathway leading to accumulation of toxic metabolite (ex : Galactosemia, Tyrosinemia type 1)
2. Involvement of cellular organelles : (Wolman's disease and Zellweger's syndrome)
3. Energy deficiency states (Mitochondrial or Cytoplasmic):(ex : fatty acid oxidation defects (FAOD) and the congenital lactic acidemias) The MLDs can present at any age, from prenatal, neonatal, infancy to adolescence and even adulthood, coinciding with the time of maximum catabolism. From the therapeutic point of view, the MLDs can be divided into four time periods e.g., neonatal age, at the time of infections, puberty and pregnancy. The diagnosis is often delayed as the symptoms may be intermittent, and in the period between episodes of decompensation, the patient may be free of clinical or biochemical abnormalities.

MLD can have varied presentations in infants and children, most common of them being: (i) organomegaly, (ii) encephalopathy due to hyperammonemia and/or primary lactic acidemia, (iii) pediatric acute liver failure (ALF), (iv) cirrhosis with or without portal hypertension, and (v) cholestatic liver disease.A high index of suspicion for MLD is important as urgent intervention such as dietary manipulation or disease-specific treatment may be life- saving.The outcome of patients undergoing liver transplantation for MLD has improved considerably over the last decade.Moreover, it is important to establish the correct diagnosis, so that appropriate genetic counselling can be offered to the family.MLD merit special attention in differential diagnosis of pediatric ALF, especially in infants and young children in whom they constitute 13- 43% of all cases .

MLDs represent 10-15% of all causes of acute liver failure in children <18 years old, with a mortality of 22-65%. In children <2-3 years of age, the percentage of acute liver failure caused by MLD rises to 33-53%.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with undiagnosed chronic hepatomegaly
2. Patients with unexplained chronic increased liver enzymes
3. Patients with undiagnosed chronic hepatomegaly or unexplained chronic increased liver enzymes and multi organ affection ( convulsions , coarse features

Exclusion Criteria:

* Patients with hepatic disorder or hepatitis with diagnosis other than metabolic ( infection ,toxic and etc …)

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Each child included in the study was subjected to the following :
  1. Detailed history : personal ,growth and developmental, perinatal ,family history and present history ( onset ,course ,duration abdominal pain , distention , jaundice , failure to thrive ,convulsions, weight loss ,stool and urine color)
  2. General examination and vital signs
  3. complete physical examination
  4. anthropometric measurements
  5. Abdominal examination ( ascitis , petechiae hepatomegaly and splenomegaly).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of metabolic liver disorders in children | Baseline
  Detect prevalence of metabolic liver disorders in children aged less than 18 years with symptoms and signs of unexplained hepatic affection admitted in Assuit university children hospital